CLINICAL TRIAL: NCT01085201
Title: Safety of Adenosine 2A Agonist Lexiscan in Children and Adults With Sickle Cell Disease
Brief Title: Adenosine 2A Agonist Lexiscan in Children and Adults With Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Boston Children's Hospital (Other); Washington University School of Medicine (Other); Medical College of Wisconsin (Other); Johns Hopkins University (Other); La Jolla Institute for Allergy & Immunology (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Principal Investigator, David G. Nathan, MD, Professor of Pediatrics, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-308; 1RC2HL101367-01 (NIH)
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-02

CONDITIONS: Sickle Cell Disease
Keywords: lexiscan
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Stage 1 (Experimental): 12-hour infusion to adults with SCD who are not having a pain crisis. THIS STAGE IS COMPLETE AND CLOSED TO ACCRUAL.
  Interventions: Drug: Lexiscan
- Stage 2 (Experimental): 24-hour infusion to adults with SCD who are not having a pain crisis. THIS STAGE IS COMPLETE AND CLOSED TO ACCRUAL.
  Interventions: Drug: Lexiscan
- Stage 3 (Experimental): 24-hour infusion to adults with SCD who are having a pain crisis. THIS STAGE IS COMPLETE AND CLOSED TO ACCRUAL.
  Interventions: Drug: Lexiscan
- Stage 4 (Experimental): 24-hour infusion to children with SCD who are having a pain crisis. THIS STAGE IS COMPLETE AFTER STUDYING 3 PATIENTS BY AGREEMENT FROM THE FDA, IRB, AND DSMB. THIS STAGE IS CLOSED TO ACCRUAL.
  Interventions: Drug: Lexiscan
- Stage 2B (Experimental): 48-hour infusion to adults with SCD who are not having a pain crisis. THIS STAGE IS COMPLETE AFTER STUDYING 3 PATIENTS BY AGREEMENT FROM THE FDA, IRB, AND DSMB. THIS STAGE IS CLOSED TO ACCRUAL.
  Interventions: Drug: Lexiscan

INTERVENTIONS:
Drug: Lexiscan — Given as an infusion

SUMMARY:
Sickle cell disease (SCD) is an inherited blood disorder that causes the red blood cells to change their shape from a round shape to a half-moon/crescent or sickled shape. People who have SCD have a different type of protein that carries oxygen in their blood (hemoglobin) then people without SCD. This different type of hemoglobin makes the red blood cells change into a crescent shape under certain conditions. Sickle-shaped cells are a problem because they often get stuck in blood vessels blocking the flow of blood, and cause inflammation and injury to the important areas in the body. Lexiscan is drug that may prevent this inflammation and injury caused by the sickle shaped cells. This drug is approved by the FDA to be used as a fast infusion during a heart stress test in people who are unable to exercise enough to put stress on their heart by making it beat faster. Lexiscan has never been studied in patients with SCD and has never been given as a long infusion.

DETAILED DESCRIPTION:
* In this research study we are looking for the highest dose of Lexiscan that can be given safely to patients with SCD. There are 4 stages to this study. Each stage will look for the highest dose that can be given safely in the following situations: Stage 1: Lexiscan will be given through a 12 hours infusion to adults with SCD who are not having a pain crisis. Stage 2: Lexiscan will be given through a 24 hour infusion to adults with SCD who are not having a pain crisis. Stage 2b: Lexiscan will be given through a 48 hour infusion to adults with SCD who are not having a pain crisis. Stage 3: Lexiscan will be given through a 24 hour infusion to adults with SCD who are having a pain crisis. Stage 4: Lexiscan will be given through a 24 hour infusion to children with SCD who are having a pain crisis. Stages 1-3 are now complete and closed to accrual. The study is now open to children ages 10-17 with SCD pain crisis (stage 4) only.
* When participants sign the consent form, they will be told what stage they will join.
* Participants in Stages 1, 2, and 2b will be given an infusion of the study drug at the time when they do not have a pain crisis. The infusion for Stage 1 participants will be 12 hours long, followed by a 6-hour observation period. The infusion for Stage 2 will be 24 hours long, followed by a 6-hour observation period. The infusion for Stage 2b will be 48 hours long, followed by a 6-hour observation period.
* Participants in Stages 3 and 4 will be given one infusion of the study drug when they are admitted to the hospital for a pain crisis. The infusion will be 24 hours long, followed by a 6-hour observation period. During the infusion, they will receive standard treatment for their pain crisis.
* Before the infusion the following procedures will be performed: Pulmonary function test (optional, Stage 1 only), blood test and vital signs.
* During the infusion the following procedures will be performed: heart rate and amount of oxygen in the blood will be monitored continuously, blood tests and blood pressure.
* During the observation period immediately following the infusion the following procedures will be performed: heart rate and amount of oxygen in the blood will be monitored continuously, blood tests, blood pressure and Pulmonary Function test (optional, Stage 1 only).

ELIGIBILITY:
Inclusion Criteria Stage I/II/IIb: (COMPLETE AND CLOSED TO ACCRUAL)

* Participants must have sickle cell anemia confirmed by hemoglobin analysis
* Participants must report that their pain is at baseline. Additionally, they cannot report an increase in dose or frequency of opioid use in the last 2 weeks prior to drug administration
* Age 21-70 years
* Participants must have the laboratory indices as outlined in the protocol
* Participants must have reliable IV access as determined by the investigator
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of the study.

Inclusion Criteria Stage III: (COMPLETE AND CLOSED TO ACCRUAL)

* Participants must have sickle cell anemia confirmed by hemoglobin analysis
* Participant is admitted to the hospital for a pain episode
* Age 21-70 years
* Participants must have the laboratory indices as outlined in the protocol
* Participants must have reliable IV access as determined by the investigator
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation

Inclusion Criteria Stage IV: (open, still accruing volunteers)

* Participants must have sickle cell disease confirmed by hemoglobin analysis
* Participant is admitted to the hospital for a pain episode
* Ages of assent (10 to 17 years at DFCI, but different depending on institution)
* Participants must have the laboratory indices as outlined in the protocol
* Participants must have reliable IV access as determined by the investigator
* Participants and parents must have the ability to understand and the willingness to sign a written informed consent and assent document
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria Stage I/II/IIb: (COMPLETE AND CLOSED TO ACCRUAL)

* Participants with a current physician diagnosis of asthma (within last 12 months), require continuous supplemental oxygen, or predicted or current use of some asthma medications.
* Participants with second- or third-degree AV block or sinus node dysfunction
* Have a history of bleeding diathesis
* Have a history of clinically overt stroke
* Have a history of severe hypertension not adequately controlled with anti-hypertensive medications
* Participants who are receiving chronic anti-coagulation or anti-platelet therapy
* Participants with a history of metastatic cancer
* Participants who have had a hospitalization or emergency room visit for any reason in the past 2 weeks
* Participants may not be receiving any other study agents or have received a study agent in the past 30 days
* Uncontrolled intercurrent illness
* Pregnant or breastfeeding women
* Participants with HIV
* Participants who have previously enrolled and received the investigational agent as part of this study
* Participants who are taking medications that may interact with the investigational agent

Exclusion Criteria Stage III: (COMPLETE AND CLOSED TO ACCRUAL)

* Participants with a current physician diagnosis of asthma (within last 12 months), require continuous supplemental oxygen, or predicted or current use of some asthma medications.
* Participants with second- or third-degree AV block or sinus node dysfunction
* Have a history of bleeding diathesis
* Have a history of clinically overt stroke
* Have a history of severe hypertension not adequately controlled with anti-hypertensive medications
* Participants who are receiving chronic anti-coagulation or anti-platelet therapy
* Participants with a history of metastatic cancer
* Participants may not be receiving any other study agents or have received a study agent in the past 30 days

Exclusion Criteria Stage IV: (open, still accruing volunteers)

* Participants with a current physician diagnosis of asthma (within last 12 months), require continuous supplemental oxygen, or predicted or current use of some asthma medications.
* Participants with second- or third-degree AV block or sinus node dysfunction
* Have a history of bleeding diathesis
* Have a history of clinically overt stroke
* Have a history of hypertension not adequately controlled with anti-hypertensive medications
* Participants who are receiving chronic anti-coagulation or anti-platelet therapy
* Participants with a history of metastatic cancer
* Participants may not be receiving any other study agents or have received a study agent in the past 30 days
* Participants with HIV
* Participants who have previously enrolled and received the investigational agent as part of this study
* Participants who are taking medications that may interact with the investigational agent

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-04; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Nathan, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - Howard University Hospital, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Childrens Hospital Boston, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Blood Center of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Field JJ, Lin G, Okam MM, Majerus E, Keefer J, Onyekwere O, Ross A, Campigotto F, Neuberg D, Linden J, Nathan DG. Sickle cell vaso-occlusion causes activation of iNKT cells that is decreased by the adenosine A2A receptor agonist regadenoson. Blood. 2013 Apr 25;121(17):3329-34. doi: 10.1182/blood-2012-11-465963. Epub 2013 Feb 1. PMID 23377438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 4/19/10 and ceased completely on 3/26/13. In Stages 1, 2 and 2b, patients were recruited from the medical clinic. For Stages 3 and 4, in which subjects were treated during a pain crisis hospitalization, patients were first informed about the study in clinic, and reminded about the study after being admitted.
Pre-assignment Details: Patients who were assigned to Stages 1, 2 or 2b, in which subjects were studied at baseline (i.e. not in pain crisis), could be excluded if they experienced a pain crisis in the interim period between enrollment and their scheduled study date.
Groups:
- Stage 1: 12-hour infusion to adults with SCD who are not having a pain crisis. THIS STAGE IS COMPLETE AND CLOSED TO ACCRUAL.
  Lexiscan : Given as an infusion
- Stage 2: 24-hour infusion to adults with SCD who are not having a pain crisis. THIS STAGE IS COMPLETE AND CLOSED TO ACCRUAL.
  Lexiscan : Given as an infusion
- Stage 2B: 48-hour infusion to adults with SCD who are not having a pain crisis. THIS STAGE IS COMPLETE AFTER STUDYING 3 PATIENTS BY AGREEMENT FROM THE FDA, IRB, AND DSMB. THIS STAGE IS CLOSED TO ACCRUAL.
  Lexiscan : Given as an infusion
- Stage 3: 24-hour infusion to adults with SCD who are having a pain crisis. THIS STAGE IS COMPLETE AND CLOSED TO ACCRUAL.
  Lexiscan : Given as an infusion
- Stage 4: 24-hour infusion to children with SCD who are having a pain crisis. THIS STAGE IS COMPLETE AFTER STUDYING 3 PATIENTS BY AGREEMENT FROM THE FDA, IRB, AND DSMB. THIS STAGE IS CLOSED TO ACCRUAL.
  Lexiscan : Given as an infusion
Period: Overall Study
Arm/Group | Stage 1 | Stage 2 | Stage 2B | Stage 3 | Stage 4
Started | 18 | 7 | 5 | 6 | 3
Completed | 15 | 6 | 3 | 6 | 3
Not Completed | 3 | 1 | 2 | 0 | 0
Not completed — Scheduling conflict | 1 | 0 | 1 | 0 | 0
Not completed — Unknown- no study drug | 2 | 0 | 0 | 0 | 0
Not completed — Fond ineligible after consent | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants was determined per protocol following a 3+3 design. In Stages 2b and 4, we received permission from the FDA, IRB, and DSMB to study only 3 subjects because we did not observe any prior DLT. One patient enrolled in Stage 2b withdrew consent during the infusion due to an unrelated toothache, and was excluded from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 | Stage 2 | Stage 2B | Stage 3 | Stage 4 | Total
Number analyzed (Participants) | 15 | 6 | 3 | 6 | 3 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 3 | 3
  Between 18 and 65 years | 15 | 6 | 3 | 6 | 0 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.71 (10.49) | 33.84 (8.75) | 23.68 (5.05) | 31.61 (6.42) | 16.77 (0.89) | 30.9 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 1 | 3 | 3 | 18
  Male | 7 | 3 | 2 | 3 | 0 | 15
Region of Enrollment [Number; unit: participants]
  United States | 15 | 6 | 3 | 6 | 3 | 33

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities as a Measure of Whether Infusional Lexiscan is Safe in Individuals With SCD.
Description: Per protocol, Lexiscan was considered "safe" if well tolerated based on number of DLTs reported. Stage 1 of the study was a 3+3 dose escalation study. Three doses were tested: 0.24 mcg/kg/hr (dose level 0), 0.6 mcg/kg/hr (dose level 1), and 1.44 mcg/kg/hr (dose level 2). Dose escalation continued until 6 participants were treated at the maximum planned dose (dose level 2). We studied a total of 15 patients in Stage 1. In Stages 2 and 3, if at least 2/3 participants tolerated the dose, an additional 3 participants were studied. We studied 6 participants in each of stages 2 and 3. In stage 2b, Lexiscan was studied for a longer (48 hr) duration in 3 participants. In stage 4, Lexiscan was studied in 3 pediatric participants.
Time Frame: 30 to 54 hours plus 30-day follow-up
Population: as for baseline characteristics
Measure: Number; unit: number of DLT
Groups:
- Stage 1 - Dose Levels 0, 1 and 2: 12-hour infusion to adults with SCD who are not having a pain crisis. THIS STAGE IS COMPLETE AND CLOSED TO ACCRUAL.
  Lexiscan : Given as an infusion
- Stage 2 - Dose Level 2: 24-hour infusion to adults with SCD who are not having a pain crisis. THIS STAGE IS COMPLETE AND CLOSED TO ACCRUAL.
  Lexiscan : Given as an infusion
- Stage 2B - Dose Level 2: 48-hour infusion to adults with SCD who are not having a pain crisis. THIS STAGE IS COMPLETE AFTER STUDYING 3 PATIENTS BY AGREEMENT FROM THE FDA, IRB, AND DSMB. THIS STAGE IS CLOSED TO ACCRUAL.
  Lexiscan : Given as an infusion
- Stage 3 - Dose Level 2: 24-hour infusion to adults with SCD who are having a pain crisis. THIS STAGE IS COMPLETE AND CLOSED TO ACCRUAL.
  Lexiscan : Given as an infusion
- Stage 4 - Dose Level 2: 24-hour infusion to children with SCD who are having a pain crisis. THIS STAGE IS COMPLETE AFTER STUDYING 3 PATIENTS BY AGREEMENT FROM THE FDA, IRB, AND DSMB. THIS STAGE IS CLOSED TO ACCRUAL.
  Lexiscan : Given as an infusion
Arm/Group | Stage 1 - Dose Levels 0, 1 and 2 | Stage 2 - Dose Level 2 | Stage 2B - Dose Level 2 | Stage 3 - Dose Level 2 | Stage 4 - Dose Level 2
Number analyzed (Participants) | 15 | 6 | 3 | 6 | 3
number of DLT | 1 | 0 | 0 | 0 | 0

2. Secondary Outcome: Percentage of Activated iNKT Cells and/or Activation Markers on iNKT Cells in Individuals With SCD.
Description: Percentage of activated iNKT cells after receiving a 24-hour infusion of Lexiscan was compared to pre-drug. iNKT cell activation was evaluated using antibodies targeting the p65 subunit of nuclear factor-kappa B (phospho-NF-kB p65). Measures are given as percentage of change in phospho-NF-kB p65 activation in iNKT cells compared to pre-drug after a 24-hour infusion. iNKT cell activation in Stages 1, 2b, and 4 was not analyzed (see analysis population description).
Time Frame: pre-drug to 54 hours
Population: The number of subjects was determined per protocol. Stage 1 was excluded as the goal was to determine the optimal markers for iNKT cells. Only 4 subjects were analyzed in Stage 2 because 24-hour samples were not obtained for 2 subjects. Stages 2b and 4 were not completely analyzed because these stages were completed early after studying 3 subjects.
Measure: Median (Standard Deviation); unit: percentage of change in activation
Arm/Group | Stage 1 - Dose Levels 0, 1 and 2 | Stage 2 - Dose Level 2 | Stage 2B - Dose Level 2 | Stage 3 - Dose Level 2 | Stage 4 - Dose Level 2
Number analyzed (Participants) | 0 | 4 | 0 | 6 | 0
percentage of change in activation |  | -3 (0.30) |  | -48 (0.30) |

3. Secondary Outcome: Pain Levels During a Vaso-occlusive Event in Children and Adults With SCD.
Description: Pain was measured using a standardized pain scale. The scale is a 10-cm visual analogue scale (10 cm-long line printed on white paper), where 0 is no pain and 10 is maximum pain. Participants were asked to indicate their pain level by marking on the line prior to each blood draw.
Time Frame: pre-drug to 54 hours
Population: The number of participants was determined per protocol following a 3+3 design. Stages 1, 2 and 2b were excluded because this outcome measure is specific to the experience of a vaso-occlusive event, which was studied in Stages 3 and 4.
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Stage 1 | Stage 2 | Stage 2B | Stage 3 | Stage 4
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 3
units on a scale |  |  |  | 5.8 (0.8) | 7.8 (1.1)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Stage 1 - Dose Levels 0, 1 and 2 | Stage 2 - Dose Level 2 | Stage 2B - Dose Level 2 | Stage 3 - Dose Level 2 | Stage 4 - Dose Level 2
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/6 | 0/3 | 1/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/15 | 0/6 | 0/3 | 0/6 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 - Dose Levels 0, 1 and 2 (N=15) | Stage 2 - Dose Level 2 (N=6) | Stage 2B - Dose Level 2 (N=3) | Stage 3 - Dose Level 2 (N=6) | Stage 4 - Dose Level 2 (N=3)
Sickle cell crisis with prolonged hospitalization - Grade 2 (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uncomplicated vaso-occlusive crisis requiring hospitalization - Grade 3 (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Rib pain, leading to hospitalization - Grade 3 (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The highest dose we examined (dose level 2, 1.44 mcg/kg/hr) may not be the maximally tolerated dose. No toxicities definitely or probably attributable to the drug occurred, so it is possible that there is a higher dose that can be tolerated safely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No